CLINICAL TRIAL: NCT06755320
Title: Comparative Study Between Airway Pressure Release Ventilation and Bi-level Positive Airway Pressure Ventilation in Acute Respiratory Distress Syndrome
Brief Title: Compare Between APRV and Bipap Ventilation in ARDS Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Ayman, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APRV versus Bipap
Record Dates: First submitted 2024-11-22; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: ARDS: Acute Respiratory Distress Syndrome; ARDS
Keywords: ARDS; APRV; BiPAP
MeSH Terms: conditions — Acute Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APRV (Other): The settings for APRV were:
  * High airway pressure (Phigh) set at the last plateau airway pressure (Pplat), not to exceed 30 cmH2O and low airway pressure (Plow) set at (5 cmH2O).
  * The release phase (Tlow) setting adjusted to terminate the peak expiratory flow rate to ≥ 50%.
  * Release frequency of 10-14 cycles/min.
  Interventions: Other: mechanical ventilation (MV)
- BiPAP (Other): The settings for BiPAP were:
  * Ti (inspiratory time) is set according to inspiratory time constant.
  * Optimum PEEP is set according to FiO2 to achieve the goal of SpO2≥90%.
  * FiO2 is set to achieve the goal of SpO2≥ 90%.
  Interventions: Other: mechanical ventilation (MV)

INTERVENTIONS:
Other: mechanical ventilation (MV) — Mechanical ventilation APRV mode ( Airway Pressure Release Ventilation )
  Arms: APRV
Other: mechanical ventilation (MV) — Mechanical Ventilation in BiPAP mode (Bi-Level Positive Airway Pressure Ventilation )
  Arms: BiPAP

SUMMARY:
To evaluate whether early use of airway pressure release ventilation would improve oxgyenation , improve lung compliance and shorten the time of mechanical ventilation compared to BIPAP ventilation in ARDS patients

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is an extremely dangerous lung condition that leads to low blood oxygen levels, and is commonly caused by sepsis, pneumonia, aspiration, and trauma. Despite great improvements in mechanical ventilation in recent years, the mortality rate of ARDS is still high. Low tidal volume ventilation (LTVV), optimum positive end-expiratory pressure, permissive hypercapnia, lung recruitment, and the prone position are common treatments for ARDS .

Lung recruitment maneuvers (LRMs) are a common element of the "open lung" approach to lung-protective ventilation. Given that atelectasis increases alveolar stress and strain during tidal ventilation, LRMs may mitigate ventilator-induced lung injury (VILI) and reduce the considerable risk of death for patients with ARDS. However, the transient application of high airway pressures may impair cardiovascular function and traumatize the pulmonary epithelium (barotrauma). Consequently, the use of LRMs is controversial .

APRV and BIPAP are modes of mechanical ventilation that allow unrestricted spontaneous breathing independent of ventilator cycling, using an active expiratory valve. Both modes are pressure-limited. Ventilation occurs via the time-cycled switching between two set pressure levels .

Bilevel positive airway pressure is a partial support mode that employs pressure-controlled, time-cycled ventilation set at two levels of continuous positive airway pressure (CPAP) with unrestricted spontaneous breathing. Which can occur at any phase of the mechanical ventilatory cycle. Bilevel positive airway pressure is able to modulate the inspiratory effort by modifying the frequency of controlled breaths .

In traditional biphasic ventilation, the inspiratory to expiratory ratio is not inverse. This ratio often distinguishes biphasic ventilation from APRV. Ventilator parameters set in this mode include the inspiratory pressure limit (Phigh), inspiratory time (Thigh), PEEP level (Plow), rate, and fraction of inspired oxgyen (FiO2). On some ventilators, pressure support may be added to augment the patient's spontaneous breaths .

Airway pressure release ventilation (APRV) is defined as a continuous positive airway pressure (CPAP) with a brief intermittent release phase based on the open lung concept; it also perfectly fits the ARDS treatment principle. Despite this, APRV has not been widely used in the past, rather only as a rescue measure for ARDS patients who are difficult to oxygenate .

APRV is a form of pressure controlled intermittent mandatory ventilation that is designed to allow unrestricted spontaneous breathing through the breath cycle, especially during Timehigh (Thigh).it is also applied using I:E ratios much greater than 1:1 or inverse ratio ventilation, usually relying on short expiratory times and gas trapping to maintain end-expiratory lung volume. APRV improve oxygenation and decrease the amount of alveolar derecruitment during the Timelow (Tlow) .

All preexisting data did not address the question for which APRV was being promoted, is that APRV should be used as initial mode of mechanical ventilation for patients with ARDS. Multiple reports and studies in animals and humans have not helped answer this question. Not only is there paucity in the number of high quality trials in humans, but there is a lack of consistency on how APRV is applied .

Over recent years, with an increased understanding of the pathophysiology of ARDS, APRV has been re-proposed to improve patient prognosis. Nevertheless, this mode is still not routinely used in ARDS patients .

Compared to the classical ventilation, APRV has been shown to provide lower peak pressure, better oxygenation, less circulatory loss, and better gas exchange without deteriorating the hemodynamic condition of the ARDS patient .

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all ARDS criteria (according to Berlin definition).
* Patients who had received endotracheal intubation and mechanical ventilation for <48h prior to inclusion.

Exclusion Criteria:

* Age below 18 years and above 65 years.
* Presence of significant chronic pulmonary disorder (chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, suppurative lung disease or diffuse alveolar hemorrhage) or documented barotrauma.
* Presence of cardiac disorder (rheumatic or ischemic heart disease).
* Presence of intracranial hypertension (suspected or confirmed).
* History of malignancies or patients on immunosuppressive drugs.
* Pregnancy or presence of neuromuscular disorder known to prolong intubation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
partial pressure of oxgyen in arterial blood | an average of 6 months
  To evaluate whether early use of airway pressure release ventilation (APRV) would improve oxygenation (as assessed by partial pressure of oxygen in the arterial blood (PaO2)).

SECONDARY OUTCOMES:
Number of days on mechanical ventilation | Up to 6 months
  recording number of days patients were on mechanical ventilation in intensive care unit (ICU )

CONTACTS AND LOCATIONS:
Overall Officials: Rana A Mohamed, MSc, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No
To ensure ultimate patients' privacy and disclosure , IPD might not be shared , but data will be available with the corresponding author on special request .

REFERENCES:
- [Background] Fredericks AS, Bunker MP, Gliga LA, Ebeling CG, Ringqvist JR, Heravi H, Manley J, Valladares J, Romito BT. Airway Pressure Release Ventilation: A Review of the Evidence, Theoretical Benefits, and Alternative Titration Strategies. Clin Med Insights Circ Respir Pulm Med. 2020 Feb 5;14:1179548420903297. doi: 10.1177/1179548420903297. eCollection 2020. PMID 32076372
- [Background] Saddy F, Moraes L, Santos CL, Oliveira GP, Cruz FF, Morales MM, Capelozzi VL, de Abreu MG, Garcia CS, Pelosi P, Rocco PR. Biphasic positive airway pressure minimizes biological impact on lung tissue in mild acute lung injury independent of etiology. Crit Care. 2013 Oct 8;17(5):R228. doi: 10.1186/cc13051. PMID 24103805
- [Background] Goligher EC, Hodgson CL, Adhikari NKJ, Meade MO, Wunsch H, Uleryk E, Gajic O, Amato MPB, Ferguson ND, Rubenfeld GD, Fan E. Lung Recruitment Maneuvers for Adult Patients with Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S304-S311. doi: 10.1513/AnnalsATS.201704-340OT. PMID 29043837
- [Background] Gallagher JJ. Alternative Modes of Mechanical Ventilation. AACN Adv Crit Care. 2018 Winter;29(4):396-404. doi: 10.4037/aacnacc2018372. PMID 30523010
- [Background] Mireles-Cabodevila E, Dugar S, Chatburn RL. APRV for ARDS: the complexities of a mode and how it affects even the best trials. J Thorac Dis. 2018 Apr;10(Suppl 9):S1058-S1063. doi: 10.21037/jtd.2018.03.156. No abstract available. PMID 29850185
- [Background] Cheng J, Ma A, Dong M, Zhou Y, Wang B, Xue Y, Wang P, Yang J, Kang Y. Does airway pressure release ventilation offer new hope for treating acute respiratory distress syndrome? J Intensive Med. 2022 Mar 28;2(4):241-248. doi: 10.1016/j.jointm.2022.02.003. eCollection 2022 Oct. PMID 36785647
- [Background] Zhong X, Wu Q, Yang H, Dong W, Wang B, Zhang Z, Liang G. Airway pressure release ventilation versus low tidal volume ventilation for patients with acute respiratory distress syndrome/acute lung injury: a meta-analysis of randomized clinical trials. Ann Transl Med. 2020 Dec;8(24):1641. doi: 10.21037/atm-20-6917. PMID 33490153
- [Background] Kucuk MP, Ozturk CE, Ilkaya NK, Kucuk AO, Ergul DF, Ulger F. The effect of preemptive airway pressure release ventilation on patients with high risk for acute respiratory distress syndrome: a randomized controlled trial. Braz J Anesthesiol. 2022 Jan-Feb;72(1):29-36. doi: 10.1016/j.bjane.2021.03.022. Epub 2021 Apr 24. PMID 33905798
- [Background] Rose L, Hawkins M. Airway pressure release ventilation and biphasic positive airway pressure: a systematic review of definitional criteria. Intensive Care Med. 2008 Oct;34(10):1766-73. doi: 10.1007/s00134-008-1216-3. Epub 2008 Jul 17. PMID 18633595